CLINICAL TRIAL: NCT06387732
Title: The Mechanisms Underlying the Antidepressant Effects of Physical Activity
Brief Title: Mechanisms Underlying Antidepressant Effects of Physical Activity
Acronym: LIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: King's College London (Other); Queen Mary University of London (Other); University of Dublin, Trinity College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 161223
Record Dates: First submitted 2023-12-15; First posted 2024-04-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Depression
Keywords: Aerobic exercise; Effort; Decision-making; Cognitive control; Dopamine; Inflammation; Motivation
MeSH Terms: conditions — Depression; Inflammation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The trial will use a single-site parallel group design with depressed participants randomised to eight weeks of either 45 minutes of aerobic exercise of moderate-to-vigorous activity (experimental group: three times per week, N=125) or 45 minutes of non-aerobic stretching/guided relaxation (control group: three times per week, N=125).
Who Masked: Participant
Masking Description: The control arm is stretching and relaxation. Prior research indicates that participants have similar efficacy expectations regarding mild stretching and aerobic exercise, which will help to improve masking. Due to the nature of the interventions, it is not possible for the participants to be masked as to the intervention they are undergoing, but all study information will be agnostic about which intervention we expect to be more effective, and all analysis will be performed by blinded staff. The trial will assess expectations and preferences about the intervention conditions, allowing for sensitivity analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): Participants will be randomised to eight weeks of 45 min aerobic exercise of moderate-to-vigorous activity (experimental group: three times per week, N=125).
  Interventions: Other: Aerobic exercise
- Stretching and relaxation (Active Comparator): Participants will be randomised to eight weeks of 45 min aerobic exercise of stretching and relaxation (control group: three times per week, N=125).
  Interventions: Other: Stretching and relaxation

INTERVENTIONS:
Other: Aerobic exercise — This will be delivered by coaches in a small group class format. Participants will complete the trial in staggered cohorts, with no more than six participants per class. Intervention activities will be tailored to each individual's own ability and fitness level.
  Arms: Aerobic exercise
Other: Stretching and relaxation — This will be delivered by coaches in a small group class format. Participants will complete the trial in staggered cohorts, with no more than six participants per class. Intervention activities will be tailored to each individual's own ability and fitness level.
  Arms: Stretching and relaxation

SUMMARY:
It is well established that any level of physical activity can help prevent and treat depression, with more strenuous activity having a greater effect. Understanding the mechanisms driving this antidepressant effect is important because it could allow exercise programmes to be made more effective, accessible, and targeted. Such knowledge could contribute to social prescribing, increasingly a priority for mental healthcare. Importantly, physical activity is highly scalable, low cost, well suited to early intervention, and has beneficial impacts on physical health co-morbidities. This trial may provide initial indications of whether there are sub-groups of depressed individuals who are particularly likely to benefit from physical activity, lead to strategies to personalise physical activity prescription based on motivational factors, and pave the way for augmentative approaches, for example combining physical activity with psychological interventions.

To date the mechanisms driving the antidepressant effects of physical activity in humans are poorly understood. Building on links between depressive symptoms, reward processing and dopamine, plus evidence from animal studies that physical activity is anti-inflammatory and boosts both dopamine and reward processing, the overarching aim of this trial is to understand the mechanisms underlying the effects of physical activity in depression, focusing on the concept of motivation.

The key objective is to conduct a randomised controlled trial (RCT) in N=250 depressed participants comparing aerobic exercise to a stretching/relaxation control condition, examining a range of mechanistic factors. The proposed trial will examine the impact of physical activity at multiple, linked potential levels of explanation: (1) immune-metabolic markers; (2) dopamine synthesis capacity; (3) activation in the brain's reward and effort processing circuitry;(4) effort-based decision making incorporating computational analysis; and (5) symptom networks based on fine-grained, daily measurements.

DETAILED DESCRIPTION:
The primary objective is to conduct a randomised controlled trial (RCT) in N=250 depressed participants comparing aerobic exercise to a stretching/relaxation control condition, examining effects on a range of potential clinical and mechanistic factors: depressive symptoms; immune-metabolic function; activation in the brain's reward and effort processing circuitry using functional magnetic resonance imaging (fMRI); cognitive tasks, focusing on reward processing; and a subset (approximately one-third) of participants will complete L-6-[18F] fluoro-3,4-dihydroxyphenylalnine (18F-DOPA) positron emission tomography (PET).

The secondary objectives are to assess: (1) the degree to which changes in the mechanistic factors are related to changes in interest-activity symptoms of depression resulting from aerobic exercise; (2) whether baseline mechanistic or clinical factors are associated with symptomatic improvement measured by symptom questionnaires following the exercise intervention; (3) whether aerobic exercise-induced changes in the brain circuits underlying cognitive control overlap with those implicated in motivation.

The trial will use an RCT design, with depressed participants randomised to eight weeks of either 45 minutes aerobic exercise of moderate-to-vigorous intensity activity (experimental group: three times per week, N=125) or 45 minutes of non-aerobic stretching/guided relaxation (control group: three times per week, N=125). The target sample size following expected attrition is N~105 per arm. Participants will complete the trial in staggered cohorts, with no more than six participants per class.

Blood and saliva samples will be taken before the intervention at baseline (between weeks -1 and 0), mid-intervention (week 3 and week 4), and post-intervention (week 9 to week 14) visits, to assess changes in immune-metabolic markers. Blood and saliva samples will also be collected at baseline and post-intervention from approximately 30 healthy controls.

Functional neuroimaging during effort-based decision-making and cognitive control will be taken at baseline and post-intervention. The same functional neuroimaging measures will also be collected at baseline and post-intervention from approximately 30 healthy controls.

Cognitive assessments will be completed online at baseline, every other week during the intervention (week 1, week 3, week 5, week 7), and post-intervention. The same cognitive assessments will also be collected at identical time-windows from approximately 30 healthy controls.

Questionnaire assessments will be completed online at baseline, every other week (week 2, week 4, week 6) and post-intervention (week 9 to 14). The same questionnaire assessments will be collected at baseline and post-intervention from approximately 30 healthy controls.

Accelerometers will measure physical activity continuously at baseline and during the intervention. Fitness testing will provide a measure of cardiovascular fitness at baseline and post-intervention visits. Daily depressive symptoms will be recorded using abbreviated scales using the Neureka smartphone app throughout the intervention. Three-monthly follow up of symptoms/cognition from baseline over six months will assess the durability of effects (week 21 and week 33).

In a subset of participants, approximately one-third of the participants will also complete a positron emission tomography (PET) scan pre-randomisation and at a visit during weeks 4-9 to 14, to assess dopamine synthesis capacity. The same PET scan will also be collected from approximately 30 healthy controls.

ELIGIBILITY:
Inclusion Criteria will include:

1. PHQ9≥12 (moderate depression).
2. Current physical activity level below 30 min moderate physical activity, once per week.
3. Fluency in English.
4. Willingness to undergo the interventions.
5. Age 18-60.
6. Willing and able to provide written informed consent.

Exclusion Criteria will include:

1. Medical contraindications to either intervention.
2. Neurological illness.
3. Past or current diagnosis of psychosis, bipolar disorder, or substance/alcohol use disorder, unless restricted to a depressive episode.
4. Unable to complete self-administered cognitive or questionnaire assessments.
5. Symptoms or cognitive impairment that would limit capacity to consent.
6. Pregnancy.
7. Regular use of anti-inflammatory medication (more than once per week).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 score | Post-intervention (week 9 to week 14)
  Depression symptoms will be measured using the Patient Health Questionnaire-9 (PHQ-9). Minimum score is 0, maximum score is 27. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Physical activity | Baseline assessment period (between weeks -1 and 0) to post-intervention (week 9 to week 14), and follow-up (weeks 21 and 33)
  Physical activity will be measured continuously by accelerometers and between baseline, post-intervention and follow-up (weeks 21 and 33) using the International Physical Activity Questionnaire (IPAQ). The minimum score is 0, and there is no maximum score. A higher score means more physical activity.
Aerobic capacity: CPET | Baseline (between weeks -1 and 0) and post-intervention (week 9 to week 14)
  Aerobic capacity will be measured by the Cardiopulmonary Exercise Test (CPET), which is a physical fitness test.
Ecological Momentary Assessment | Baseline assessment period (between weeks -1 and 0) to post-intervention (week 9 to week 14)
  Brief daily depressive symptoms will be recorded throughout the intervention, using abbreviated scales, through the Neureka smartphone app. Minimum score per item is -3, maximum score per item is 3. Higher scores mean a worse outcome.
Inflammatory response (cytokines) | Baseline (between weeks -1 and 0), mid-intervention (week 3 or week 4), and post-intervention (week 9 to week 14)
  Inflammatory cytokines (pg/mL) will assess changes in inflammatory responses.
Inflammatory response (genetic markers) | Baseline (between weeks -1 and 0), mid-intervention (week 3 or week 4), and post-intervention (week 9 to week 14)
  Transcriptional markers (fold change) will assess changes in inflammatory responses.
Inflammatory response (flow cytometry immunophenotype) | Baseline (between weeks -1 and 0), mid-intervention (week 3 or week 4), and post-intervention (week 9 to week 14)
  Flow cytometry immunophenotype (% cells) will assess changes in inflammatory responses.
Neuroendocrine system | Baseline (between weeks -1 and 0), mid-intervention (week 3 or week 4), and post-intervention (week 9 to week 14)
  Cortisol over the day (pg/mL) will assess changes in the neuroendocrine system.
Metabolic function | Baseline (between weeks -1 and 0), mid-intervention (week 3 or week 4), and post-intervention (week 9 to week 14)
  Metabolic blood markers (mg/dl) will assess changes in metabolic function.
Dopamine synthesis capacity | Baseline (between weeks -1 and 0) and post-intervention (week 4-9 to week 14)
  In a subset of participants, dopamine synthesis capacity measured by 18F-DOPA PET will be taken.
Functional magnetic resonance imaging (fMRI) during cognitive tasks | Baseline (between weeks -1 and 0) and post-intervention (week 9 to week 14)
  Participants will complete effort-based decision making and cognitive control tasks during fMRI.
Online cognitive tasks | During every other week of the intervention (weeks -1/0, week 1, week 3, week 5, week 7, week 9 to week 14)
  Participants will complete online cognitive tests of effort-based decision-making and cognitive control, alongside other tests of reward processing.
Depression symptoms | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6)
  Depression symptoms will be measured by the Patient Health Questionnaire-9 (PHQ-9). Minimum score is 0, maximum score is 27. Higher scores mean a worse outcome.
Anxiety (GAD7 score) | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6, week 9 to week 14)
  Anxiety will be measured by the Generalised Anxiety Disorder Assessment (GAD7). Minimum score is 0, maximum score is 21. Higher scores mean a worse outcome.
Anxiety (STAI score) | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6, week 9 to week 14)
  Anxiety will be measured by the State-Trait Anxiety Inventory (STAI). Minimum score is 20, maximum score is 80. Higher scores mean a worse outcome.
Anhedonia (SHAPS score) | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6, week 9 to week 14)
  Anhedonia will be measured by the Snaith-Hamilton Pleasure Scale (SHAPS). Minimum score is 14, maximum score is 56. Higher scores mean a better outcome.
Anhedonia (DARS score) | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6, week 9 to week 14)
  Anhedonia will be measured by the Dimensional Anhedonia Rating Scale (DARS). Minimum score is 0, maximum score is 68. Higher scores mean a better outcome.
Apathy | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6, week 9 to week 14)
  Apathy will be measured by the Apathy Evaluation Scale (AES). Minimum score is 18, maximum score is 72. Higher scores mean a worse outcome.
Fatigue | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6, week 9 to week 14)
  Fatigue will be measured by the Fatigue Severity Scale (FSS). Minimum score is 9, maximum score is 63. Higher scores mean a worse outcome.
Cognitive impairment | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6, week 9 to week 14)
  Cognitive impairment will be measured by the British Columbia Cognitive Complaints Inventory (BC-CCI). Minimum score is 0, maximum score is 18. Higher scores mean a worse outcome.
Self-efficacy | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6, week 9 to week 14)
  Self-efficacy will be measured by the General Self-Efficacy Scale (GSES). Minimum score is 8, maximum score is 40. Higher scores mean a better outcome.
Self-esteem | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6, week 9 to week 14)
  Self-esteem will be measured by the Single-Item Self-Esteem Scale (SISES). Minimum score is 1, maximum score is 7. Higher scores mean a better outcome.
Sleep quality | During every other week of the intervention (weeks -1/0, week 2, week 4, week 6, week 9 to week 14)
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI). Minimum score is 0, maximum score is 21. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Roiser, PhD, Principal Investigator — University College, London
Locations (1):
- Institute of Cognitive Neuroscience, University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified questionnaire, cognitive, activity, EMA and immune-metabolic data through online repositories. We will share de-identified MRI and PET data on request through managed access agreements.
Time Frame: Anonymised data will be available for sharing after publication of the trial results. Data will be available indefinitely.